CLINICAL TRIAL: NCT06432582
Title: Assessment of a hepatomiR Cut-off for Predicting Specific Hepatic Decompensation Events in Advanced Chronic Liver Disease
Brief Title: hepatomiR cACLD Study
Status: Recruiting | Type: Observational
Sponsor: Karl Landsteiner University of Health Sciences (Other)
Collaborators: University Hospital St. Polten (Other)
Responsible Party: Sponsor
Other Study IDs: UKStP_hepatomiR_cACLD
Record Dates: First submitted 2024-05-16; First posted 2024-05-29 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Chronic Liver Disease and Cirrhosis; Chronic Liver Disease; Portal Hypertension
Keywords: hepatomiR; micro-RNA; hepatic decompensation; ACLD
MeSH Terms: conditions — Fibrosis; Hypertension, Portal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- cACLD: Patients with compensated advanced chronic liver disease (cACLD) regardless of etiology
  Interventions: Diagnostic Test: hepatomiR

INTERVENTIONS:
Diagnostic Test: hepatomiR — hepatomiR is a CE-certified test intended for gauging liver-related outcomes. It quantifies the levels of hsa-miR-122-5p, hsa-miR-192-5p, and hsa-miR-151a-5p in human plasma samples. A proprietary algorithm is then used to compute a liver function score (hepatomiR p-score).

SUMMARY:
This study looks to gather data on hepatomiR, a CE-certified test already intended for gauging liver-related outcomes, in order to define a cut-off regarding specific decompensation events (ascites, variceal hemorrhage, hepatic encephalopathy) in chronic liver disease (CLD). Based on these data, it is aimed to advance the current understanding of factors driving decompensation, with potential repercussions for future risk management and therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Chronic liver disease (more than 6 months)
* LSM ≥ 10 kPa
* Outpatient at the Clinical Department of Internal Medicine II, University Hospital St. Pölten
* Signed patient consent form

Exclusion Criteria:

* Age older than 18 years
* Pregnancy
* Primary hepatic malignancy (hepatocellular carcinoma, cholangiocarcinoma) with portal invasion and/or extrahepatic spread

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is made up of patients with compensated advanced chronic liver disease (cACLD) regardless of etiology; cACLD will be defined as per the Baveno VII consensus (LSM values: ≥ 10 kPa ACLD, less than 10 kPa non-ACLD).
Sampling Method: Non-Probability Sample
Enrollment: 156 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Occurrence of any hepatic decompensation event (per patient) | 12 months
  Any (further) hepatic decompensation event (compound endpoint; Baveno VII definition; ascites, variceal bleeding, hepatic encephalopathy)

SECONDARY OUTCOMES:
Number and type of individual decompensation events (per patient) | 12 months
Number of hospital admissions (per patient) | 12 months
Number of acute on chronic liver failure events (per patient) | 12 months
  EF-CLIF (European Association for the Study of the Liver - Chronic Liver Failure) definition, CLIF-C (chronic liver failure score) ACLF (acute on chronic liver failure) grading
Number of ICU (intensive care unit) admissions (per patient) | 12 months
Development of hepatocellular cancer or cholangiocarcinoma (per patient) | 12 months
Number of deaths | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Maieron, PD Dr., Principal Investigator — Karl Landsteiner University of Health Sciences
Locations (1):
- University Hospital St. Pölten, Sankt Pölten, Lower Austria, Austria

IPD SHARING:
Plan to Share IPD: No